CLINICAL TRIAL: NCT03926182
Title: A Randomized, Open Label, Single Center, Crossover Study to Determine the Effect of Food on the Pharmacokinetics of Single Oral Doses of Alflutinib Mesylate Tablets (AST2818) in Healthy Male Volunteers in the Fasted State or Following a High Fat Meal
Brief Title: Study to Determine the Effect of Food on the Blood Levels of AST2818 Following Single Oral Doses in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20190120
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted AST2818 tablets following a period of fasting (Experimental)
  Interventions: Drug: AST2818 Tablets
- High-fat meal AST2818 tablets following a high-fat meal (Experimental)
  Interventions: Drug: AST2818 Tablets

INTERVENTIONS:
Drug: AST2818 Tablets — AST2818 Tablets: Period 1 Fasted from 10 hours prior to dosing with 80 mg AST2818 tablet (p o, once) and 4 hours after dosing on day 1. Period 2 Allocated high-fat meal prior to dosing with 80 mg AST2818 tablet (p o, once) and fasted 4 hours after dosing on day 1.
  Arms: Fasted AST2818 tablets following a period of fasting
Drug: AST2818 Tablets — AST2818 Tablets: Period 1 allocated high-fat meal prior to dosing with 80 mg AST2818 tablet (p o, once) and fasted 4 hours after dosing on day 1. Period 2 fasted from 10 hours prior to dosing with 80 mg AST2818 tablet (p o, once)and 4 hours after dosing on day 1.
  Arms: High-fat meal AST2818 tablets following a high-fat meal

SUMMARY:
To assess the Effect of Food on the Blood Levels of AST2818 Following Single Oral Doses in Healthy Male Volunteers in Fasting State or Following a High Fat Meal

DETAILED DESCRIPTION:
This is a single center, randomized, open label, single dose, two periods crossover study in healthy male volunteers. The volunteers will be randomly distributed into two groups (fasted-fed and fed-fasted groups). Any volunteer will be administrated once in each treatment period, the interval time of two treatment periods is 22 days (the interval time is no longer than 30 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male must be ≥ 18 and ≤ 55 years of age.
2. Bodyweight of male must be ≥50.0kg and ≤80kg, and the Body Mass Index must be ≥19.0 and ≤26.0 kg/m2.
3. The results of previous medical history in screening period, physical examination, vital signs, blood and urine routine examination, blood biochemistry, chest X-ray and ECG should compliance with the clinical protocol, or they will be recognized as non-clinical signs (NCS) if beyond the regulated range.
4. The results of echocardiographic examination should meet the criteria that the LVEF value measured by biplane Simpson method was ≥ 50%.
5. The participants must have no birthing plan and agree to take adequate non-drug contraceptive measures within the study to 4 months after the last drug treatment.
6. The participants have good communications with investigators, understand and comply with all requirements and fully understand and sign the informed consent form.

Exclusion Criteria:

1. The participants have history of chronic disease and serious illness in vascular system, blood system, urinary system, respiratory system, digestive system, nervous system, skin system and psychiatric disorders, any conditions and illness threat to the health of participants, and the history of hereditary disease.
2. The participants have history of similar drug, allergy history to similar drug, allergic disorders and allergic constitution.
3. The participants having history of drug abuse，opioid and tranquillizer， drug addicts, or drug screening for someone was positive.
4. Resting corrected electrocardiogram QT interval using Fridericia's correction factor (QTcF) >470 msec within screening period.
5. Any factors that increase the risk of prolonging QTc and abnormality in heart rate, i.e., heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome or unreasonable sudden death at age smaller than 40 in first-degree relatives, administrating any combined medicines that possibly prolong QT interval
6. Severe disease of respiratory system, i.e., interstitial lung disease and severe asthma, etc.
7. Severe disease of ophthalmic system, e.g., corneal diseases;
8. The participants have severe infection, severe trauma or major surgery within 1 year before screening;
9. The participants have history of alcohol abuse (it was defined as that the daily alcohol consumption was higher than the following criteria: the weekly alcohol consumption was higher than 14 units of alcohol (1 unit= 360 ml beers/45 ml liquor containing 40% alcohol/150ml grape wine) 6 months prior to screening period, positive results of alcohol breath test and the volunteers who cannot give up drinking during study.
10. The participants who smoked daily >5 sticks of cigarette 3 months prior to first dose or cannot give up smoking during study.
11. The participants who have blood donation or excessive bleeding(>200ml) 3 months prior to first dose, and planned to donate blood or blood constituent.
12. The participants who were taking any prescription medicine、CYP3A4 inducers/inhibitors within 1 month prior to first dose; any OTC, health care products (including vitamins), traditional chinese medicine within 2 weeks prior to screening period.
13. The participants who participated other clinical trials and took the investigational drug 3 months prior to first dose.
14. The participants who have positive test result in HBsAg, Anti-HCV, Anti-HIV and TPPA.
15. Any condition affecting the drug taking, or affecting the oral absorption, include any kind of severe chronic gastroenteropathy, history of gastrointestinal resection or surgery, uncontrollable nausea or vomit, disability in swallowing.
16. The participants who have history of needlesickness and blood phobia, and those with severe bleeding tendency.
17. The participants who cannot comply with the roles of unified diet.
18. The participants who cannot tolerate blood collection through venipuncture.
19. The participants who have chronic overconsumption (> 8 cup one day, 1 cup=250 ml) of tea, coffee, and the drink with caffeine; or intake food or drink consist of any caffeine (i.e., coffee, strong tea, and chocolate );
20. Any intake of drink or food, enriched in xanthine and grapefruit, that could affect the drug's absorption, distribution, metabolism and excretion.
21. Any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Cmax of AST2818 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST2818 by assessment of maximum plasma AST2818 concentration.
AUC(0-t) of AST2818 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST2818 by assessment of area under the plasma concentration time curve from zero to appointed time
Tmax of AST2818 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST2818 by assessment of time to Cmax.

SECONDARY OUTCOMES:
Cmax of AST5902 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST5902 (metabolite to AST2818) by assessment of maximum plasma AST5902 concentration.
AUC(0-t) of AST5902 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST5902 (metabolite to AST2818) by assessment of area under the plasma
Tmax of AST5902 | Blood samples collected on Day 1 at 0.5 hour of pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post AST2818 dose in each period of two groups.
  Pharmacokinetics of AST5902 (metabolite to AST2818) by assessment of time to Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Tumor Hospital, Changsha, Hunan, China